CLINICAL TRIAL: NCT01935700
Title: Evaluation the Potential of Colchicine for the Palliative Management of Hepatocellular Carcinoma Patients With Distant Metastasis or Large Vessel Invasion
Brief Title: Effect of Colchicine for the Palliative Management of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Zu-Yau Lin, professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-04-03(I)
Record Dates: First submitted 2013-08-24; First posted 2013-09-05 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma; Metastasis; Invasion
Keywords: hepatocellular carcinoma; colchicine
MeSH Terms: conditions — Carcinoma, Hepatocellular; Neoplasm Metastasis | interventions — Colchicine; Colicins

STUDY DESIGN:
Intervention Model Description: opeo labeled
Oversight: Data Monitoring Committee: No

ARMS (1):
- colchicine treated patients (Experimental): 2 tablets (0.5 mg/tablet) of colchicine three times per day (after breakfast, lunch and dinner); continue 4 days and stop for 3 days (1 cycle); repeat this cycle until patients quit this trial
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — Adjustment the dosage of colchicine during study:
  The colchicine dosage will be changed when the hepatic reserved function of the participant changes from Child A to B according as following: 2 tablets after breakfast, 1 tablet after lunch and 2 tablets after dinner; continue 4 days and stop for 3 days (1 cycle); repeat this cycle until patients quit this trial. If the hepatic reserved function of the participant changes to Child C, colchicine will be stopped and participant receives regular follow-up only.If participant suffers from severe diarrhea, colchicine will be temporarily stopped. When the symptom of diarrhea subsides, colchicine will be given again but the dose will be reduced 0.5 mg/day.
  Other Names: Colicine, Tunfon and others, Drugbank Accession Number DB01394, PubChem CID 6167, CAS Registry Number: 64-86-8

SUMMARY:
This trial is to evaluate the potential of colchicine for the palliative management of hepatocellular carcinoma patients with distant metastasis or large vessel invasion using the Department of Health R.O.C. approved doses and methods of administration.

DETAILED DESCRIPTION:
Dosing schedule: 2 tablets (1 mg) three times per day (after breakfast, lunch and dinner); continue 4 days and stop for 3 days (1 cycle)

Adjustment the dosage of colchicine during study:

1. The colchicine dosage will be changed when the hepatic reserved function of the participant changes from Child A to B according to the following rules.

   1. 2 tablets after breakfast, 1 tablet after lunch and 2 tablets after dinner; continue 4 days and stop for 3 days (1 cycle); repeat this cycle until patients quit this trial
   2. If the hepatic reserved function of the participant returns to Child A, The dosage for Child A will be restored.
   3. If the hepatic reserved function of the participant changes to Child C, colchicine will be stopped and participant receives regular follow-up only.
2. If participant suffers from severe diarrhea, colchicine will be temporarily stopped. When the symptom of diarrhea subsides, colchicine will be given again according to the following rules.

   1. For participant receives﹝2 tablets after breakfast, 2 tablet after lunch and 2 tablets after dinner﹞, the dosage of colchicine will be changes to﹝2 tablets after breakfast, 1 tablet after lunch and 2 tablets after dinner﹞.

      If diarrhea attacks again, the dosage of colchicine will be changes to﹝2 tablets after breakfast and 2 tablets after dinner﹞.

      If diarrhea attacks again, the dosage of colchicine will be changes to﹝2 tablets after breakfast, 1 tablet after dinner﹞.

      If diarrhea also attacks again, colchicine will be stopped and participant receives regular follow-up only.
   2. For participant receives﹝2 tablets after breakfast, 1 tablet after lunch and 2 tablets after dinner﹞, the dosage of colchicine will be changes to﹝2 tablets after breakfast and 2 tablets after dinner﹞.

   If diarrhea attacks again, the dosage of colchicine will be changes to﹝2 tablets after breakfast, 1 tablet after dinner﹞.

   If diarrhea also attacks again, colchicine will be stopped and participant receives regular follow-up only.
3. If the participant has one of the following conditions, colchicine will be temporarily stopped. When the condition of the participant improves, colchicine will be given again after the judgment from the doctor of the research team. For participants unable to receive colchicine again, they will receive regular follow-up only.

   1. There are life-threatening hemorrhage including gastrointestinal hemorrhage and hemorrhage from other vital organs such as lungs or brain.
   2. . There are life-threatening bacterial, fungal or viral infection (not included hepatitis B and C virus).
   3. . Patient has serum creatinine level > 1.5 mg/dL.
   4. . Patient has white blood cell count < 1500/µL, platelet count < 30000/µL or hemoglobin < 9.0 gm/dL after medication.
   5. The research team decides that the participant is not suitable to continue the study caused by abnormality of any vital organ or severe side effects caused by the study.
4. Colchicine will be temporarily stopped one day before transcatheter arterial chemoembolization until participant has body temperature < 38 ℃, same hepatic reserved function as before, and serum creatinine level < 1.5 mg/d after embolization.

Follow-up procedures and items for the participants to co-operate:

All participants will be followed according to the guide line of the National Health Council and the clinical practice in the treatment of hepatocellular carcinoma. Contrasted-enhanced computed tomography or magnetic resonance imaging will be performed within every 3 to 4 months. Serum alpha-fetoprotein will be determined at least one session within every 2 to 3 months in patients with elevated serum alpha-fetoprotein levels. The hepatic and renal function will be determined at least one session every month. The participants are asked to visit our outpatient clinic at least one session every month.

ELIGIBILITY:
Inclusion Criteria:

1. . Patient has at least one of the following criteria: (1) positive for hepatocellular carcinoma evidenced by cytology or pathology, (2) serum alpha-fetoprotein level > 400 ng/mL and has evidence of hepatocellular carcinoma provided by contrast-enhanced computed tomography or magnetic resonance imaging.
2. . Contrast-enhanced computed tomography or magnetic resonance imaging has evidence of distant metastasis or large vessel invasion caused by hepatocellular carcinoma.
3. . Patient has Child A hepatic reserved function

Exclusion Criteria:

1. . There are life-threatening hemorrhage including gastrointestinal hemorrhage and hemorrhage from other vital organs such as lungs or brain.
2. . There are life-threatening bacterial, fungal or viral infection (not included hepatitis B and C virus).
3. . Patient has serum creatinine level > 1.5 mg/dL.
4. . Patient must receive long-term medication of statin or fibrates drugs and these medications can not be changed.
5. . Patient has white blood cell count < 1500/µL, platelet count < 30000/µL or hemoglobin < 9.0 gm/dL after medication.
6. . Pregnant woman or plan to be a pregnant woman
7. . allergy to colchicine or has history of severe side effects caused by colchicine
8. . Patient has received systemic chemotherapy within 2 months before enrollment or plans to receive systemic chemotherapy in the future.
9. . Patient is under or plans to receive Nexavar or other clinical trial testing drug.
10. . Patient has severe malfunction of vital organs and can not participate in this study justified by the doctor in this research team.
11. . Patient is under or plans to receive Chinese traditional medicine or herb drugs.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zu Y Lin, MS, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Lin ZY, Wu CC, Chuang YH, Chuang WL. Anti-cancer mechanisms of clinically acceptable colchicine concentrations on hepatocellular carcinoma. Life Sci. 2013 Sep 3;93(8):323-8. doi: 10.1016/j.lfs.2013.07.002. Epub 2013 Jul 16. PMID 23871804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from 2013-6-6 to 2019-5-31 in Kaohsiung Medical University Hospital total 15 participants were included for screening, one screening failure, 14 participants received colchicine management
Pre-assignment Details: one screening failure dut to active gastrointestinal hemorrhage
Groups:
- Colchicine Treated Patients: The dosing schedule started from 1 mg three times per day after meal for 4 days and stopped for the following 3 days (1 cycle). This cycle was repeated till the participant quitted this trial.
  Adjustment of colchicine dosage during study:
  1. The colchicine dosage was changed when the hepatic reserved function of the participant changed from Child A to B or C according to the following rules.
     1. Total daily dose reduced to 2.5 mg (1mg morning, 0.5 mg afternoon, 1 mg night) for participant with Child class B.
     2. If the participant changed to Child class C, colchicine will be stopped and participant received regular follow-up only.
  2. Colchicine was temporarily stopped in participant suffered from diarrhea and was started again with reducing daily total dose of 0.5 mg.
  3. Colchicine was temporarily stopped when the participant fitted any of the exclusion criteria during the study, and was given again after the fitted exclusion criterion was eliminated.
- Sorafenib Treated Group: This group was originated from review of hepatocellular carcinoma patients (from January 1, 2014 to May 31, 2019) with the same condition as this trial selected participants and treated by sorafenib for more than 2 months by the research team.
Period: Overall Study
Arm/Group | Colchicine Treated Patients | Sorafenib Treated Group
Started | 14 | 86
Completed (The participant received more than 8 courses of colchicine management.) | 9 | 86
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 4 | 0

BASELINE CHARACTERISTICS:
Population: The participant received more than 8 courses of colchicine management.
Groups:
- Colchicine Treated Patients: This group included participants receiving total daily colchicine dose equal or larger than 1.5 mg for more than 8 cycles (28 days).
- Total: Total of all reporting groups
Arm/Group | Colchicine Treated Patients | Sorafenib Treated Group | Total
Number analyzed (Participants) | 9 | 86 | 95
Age, Continuous [Median (Full Range); unit: years] | 60 [53 to 77] | 62 [26 to 83] | 62 [26 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 1 | 19 | 20
  sex: Male | 8 | 67 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Only Taiwanese were included.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 9 | 86 | 95
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Only Taiwanese were included.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 9 | 86 | 95
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 0 | 0 | 0
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — open labeled phase II for AJCC TNM IIIB to IVB hepatocellular carcinoma patient
  Participants
    Taiwan | 9 | 86 | 95

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: The overall survival of the participants calculated from the date of enrollment to the date of death will be compared with the control group with the same TNM and the Barcelona Clinic Liver Cancer (BCLC) staging collected from 2005/1/1 to the end of this study. The overall survival of the control group was calculated from the date of receiving sorafenib treatment to the date of death.
Time Frame: up to 72 months
Population: median survival
Measure: Median (Full Range); unit: days
Groups:
- Colchicine Group: Participant received more than 8 courses of colchicine management.
- Sorafenib Treated Group: The control group was originated from review of hepatocellular carcinoma patients (from January 1, 2014 to May 31, 2019) with the same condition as this trial selected participants and treated by sorafenib for more than 2 months by the research team.
Arm/Group | Colchicine Group | Sorafenib Treated Group
Number analyzed (Participants) | 9 | 86
days | 333 [123 to 1000] | 290 [74 to 1560]
Statistical Analysis 1: Comparison: Colchicine Group vs Sorafenib Treated Group; Test type: Non-Inferiority — Non-inferiority was defined as no statistically significant difference (P value > 0.05) in median survival between the colchicine group and the sorafenib treated group; p = 0.4593, Mann-Whitney U test
Statistical Analysis 2: Comparison: Colchicine Group vs Sorafenib Treated Group; Test type: Non-Inferiority — Non-inferiority was defined as no statistically significant difference (P value > 0.05) in survival between the colchicine group and the sorafenib treated group; p = 0.3290, Log Rank

2. Secondary Outcome: Grade III Severe Adverse Events
Description: The type and frequency of grade III severe adverse events based on the Common Terminology Criteria for Adverse Events (CTCAE) noted during the study period.
Time Frame: up to 72 months
Measure: Number; unit: participants
Groups:
- Colchicine Group: This included the events occured after the participant signed the inform consent.
Arm/Group | Colchicine Group | Sorafenib Treated Group
Number analyzed (Participants) | 14 | 86
participants
  Diarrhea | 1 | 4
  Anorexia | 1 | 0
  Biliary tract obstruction | 2 | 0
  Abdominal pain | 1 | 3
  Hypoglycemia | 1 | 0
  Pneumonia | 3 | 4
  Peritonitis | 2 | 1
  Cholangitis | 2 | 2
  Sepsis | 0 | 2
  Skin rash | 0 | 1
  Palmar-plantar erythrodysesthesia syndrome | 0 | 4
  Hypertension | 0 | 2
  Hemorrhage | 0 | 8
  Hyperglycemia | 0 | 1
  Hypocalcemia | 0 | 1
  Pleural effusion | 0 | 1
Statistical Analysis 1: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of pneumonia between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.0552, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 2: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of biliary tract obstruction between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.0184, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 3: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of cholangitis between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.0931, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 4: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of peritonitis between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.0506, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 5: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of sepsis between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 6: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of diarrhea between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.5374, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 7: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of anorexia between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.14, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 8: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of abdominal pain between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.4584, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 9: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of skin rash between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 10: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of palmar-plantar erythrodysesthesia syndrome between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 11: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of hypertension between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 12: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of hemorrhage between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.5958, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 13: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of hypoglycemia between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 0.14, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 14: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of hyperglycemia between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 15: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of hypocalcemia between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05
Statistical Analysis 16: Comparison: Colchicine Group vs Sorafenib Treated Group; Comparison the incidence of grade III adverse event of pleural effusion between two groups; Test type: Equivalence — The threshold for statistically significant difference in incidence was P = 0.05; p = 1, Fisher Exact — The threshold for statistically significant difference in incidence was P = 0.05

ADVERSE EVENTS:
Time Frame: up to 72 months
Description: The adverse event for diarrhea was defined as watery or not-formed stool passage for more than 3 times per day.
Groups:
- Colchicine Group: 2 tablets (0.5 mg/tablet) of colchicine three times per day (after breakfast, lunch and dinner); continue 4 days and stop for 3 days (1 cycle); repeat this cycle until patients quit this trial
  Colchicine: Adjustment the dosage of colchicine during study:
  The colchicine dosage will be changed when the hepatic reserved function of the participant changes from Child A to B according as following: 2 tablets after breakfast, 1 tablet after lunch and 2 tablets after dinner; continue 4 days and stop for 3 days (1 cycle); repeat this cycle until patients quit this trial. If the hepatic reserved function of the participant changes to Child C, colchicine will be stopped and participant receives regular follow-up only.If participant suffers from severe diarrhea, colchicine will be temporarily stopped. When the symptom of diarrhea subsides, colchicine will be given again but the dose will be reduced 0.5 mg/day.
Arm/Group | Colchicine Group | Sorafenib Treated Group
All-Cause Mortality (participants affected / at risk) | 13/14 | 81/86
Serious Adverse Events (participants affected / at risk) | 10/14 | 33/86
Other Adverse Events (participants affected / at risk) | 14/14 | 74/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Group (N=14) | Sorafenib Treated Group (N=86)
diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (4)
anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0)
biliary tract obstruction (Hepatobiliary disorders) | 2 (3) | 0 (0) — caused by previous irradiation therapy
abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
pneumonia (Infections and infestations) | 3 (3) | 4 (5)
peritonotis (Infections and infestations) | 2 (2) | 1 (1)
Cholangitis (Infections and infestations) | 2 (3) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 8 (11)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colchicine Group (N=14) | Sorafenib Treated Group (N=86)
diarrhea (Gastrointestinal disorders) | 14 (40) | 36 (83) — grade I or II
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 31 (58) — grade I or II
Nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 15 (28) — grade I or II
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 14 (18) — grade I or II
Hypertension (Vascular disorders) | 0 (0) | 13 (17) — grade I or II
Skin rash (Skin and subcutaneous tissue disorders) | 0 (0) | 13 (29) — grade I or II
Oral mucositis (Gastrointestinal disorders) | 0 (0) | 5 (6) — grade I or II

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT01935700/Prot_SAP_000.pdf